CLINICAL TRIAL: NCT04748692
Title: Effectiveness of Exercise Therapy Versus Spinal Manual Therapy in Patients With Patellofemoral Pain Syndrome: Medium Term Follow-up Results of a Randomised Controlled Trial
Brief Title: Effectiveness of Exercise Therapy Versus Spinal Manual Therapy in Patients With PFPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Scafoglieri Aldo, Prof. dr. Aldo Scafoglieri, Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL57207.096.16
Record Dates: First submitted 2021-01-28; First posted 2021-02-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: effectiveness; exercise therapy; manipulative therapy; medium term; randimozed controlled trial
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial with a follow-up of 6 weeks. Patients with PFPS will be randomly assigned to one of two intervention groups using an online computer-based pseudo-random number generator on which the numbers were generated by use of a complex algorithm (seeded by the computer's clock). The flow diagram of the progress through the phases of the parallel randomised trial of both intervention groups (that is, enrolment, allocation, follow-up, and data analysis) follows the PRISMA statement.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The allocation of the patients to their treatment group will be concealed from the researcher that assesses the outcome measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local exercise therapy (Experimental): The local exercise therapy group focused on strengthening knee and hip muscles three times a week for 6 weeks. Once a week, patients trained with the support of a physiotherapist. The physiotherapist gradually increased the intensity of the exercises improving muscle endurance. The exercises were supplemented with mobilisations of the patellofemoral joint. Twice a week, patients trained at home following a prescribed exercise program writing down their work-out in an exercise journal.
  Interventions: Procedure: Local exercise therapy
- Spinal manual therapy (Experimental): The spinal manual therapy group was treated one a week for 6 weeks. Before the first intervention an experienced manual therapist performed a clinical examination of the lower back, SIJ, hip and knee. Anatomical maps showing innervation areas of spinal nerve roots were used to explain the regional interdependence model in the treatment of anterior knee pain. Manual therapy treatment included manipulations of the thoracolumbar (T12-L3) region or SIJ as well as hip joint. Manipulation was conducted if a restriction of range of motion was found in any of the regions. Patients were also asked to do home exercises focusing on mobilizing the thoracolumbar region and to write down their performance in an exercise journal.
  Interventions: Procedure: Spinal manual therapy

INTERVENTIONS:
Procedure: Local exercise therapy — The local exercise therapy group will focus on strengthening knee and hip muscles three times a week for 6 weeks. Once a week, patients will train with the support of a physiotherapist. The physiotherapist gradually increases the intensity of the exercises improving muscle endurance. The exercises will be supplemented with mobilisations of the patellofemoral joint. Twice a week, patients train at home following a prescribed exercise program writing down their work-out in an exercise journal.
  Arms: Local exercise therapy
Procedure: Spinal manual therapy — The spinal manual therapy group will be treated one a week for 6 weeks. Before the first intervention an experienced manual therapist performed a clinical examination of the lower back, SIJ, hip and knee. Anatomical maps showing innervation areas of spinal nerve roots will be used to explain the regional interdependence model in the treatment of anterior knee pain. Manual therapy treatment will include manipulations of the thoracolumbar (T12-L3) region or SIJ as well as hip joint. Manipulation will be conducted if a restriction of range of motion will be found in any of the regions. Patients will also be asked to do home exercises focusing on mobilizing the thoracolumbar region and to write down their performance in an exercise journal.
  Arms: Spinal manual therapy

SUMMARY:
Preliminary results of a pilot study in The Bergman Clinic Naarden (NL) show that a local exercise therapy group may decrease pain by 30% on the visual analogue scale (VAS) after 6 weeks. A reduction of 50% on the VAS was realized in a spinal manual therapy group. Therefore, the aim of this study is to compare the effectiveness of local exercise therapy versus spinal manual therapy in patients with PFPS after 6 weeks of intervention and at 6 weeks of follow-up. To the knowledge of the authors, the clinical effectiveness of spinal manual manipulations on pain, function and strength has not been investigated in the medium term.

DETAILED DESCRIPTION:
Interventions

The local exercise therapy group will focus on strengthening knee and hip muscles three times a week for 6 weeks. Once a week, patients will train with the support of a physiotherapist. The physiotherapist gradually increases the intensity of the exercises improving muscle endurance. The exercises will be supplemented with mobilisations of the patellofemoral joint. Twice a week, patients train at home following a prescribed exercise program writing down their work-out in an exercise journal.

The spinal manual therapy group will be treated one a week for 6 weeks. Before the first intervention an experienced manual therapist performed a clinical examination of the lower back, SIJ, hip and knee. Anatomical maps showing innervation areas of spinal nerve roots will be used to explain the regional interdependence model in the treatment of anterior knee pain. Manual therapy treatment will include manipulations of the thoracolumbar (T12-L3) region or SIJ as well as hip joint. Manipulation will be conducted if a restriction of range of motion will be found in any of the regions. Patients will also be asked to do home exercises focusing on mobilizing the thoracolumbar region and to write down their performance in an exercise journal.

The allocation of the patients to their treatment group will be concealed from the researcher that assesses the outcome measures.

Outcome measures The following baseline characteristics will be self-reported: age (in years), weight (in kg), height (in cm), duration of symptoms (in months), weekly participation in sport (yes/no), previously receiving exercise therapy treatment for the knee (yes/no). Patellofemoral chondral lesions will be graded using the Kellgren and Lawrence system for classification of osteoarthritis (grade 0 = definite absence of X-ray changes of osteoarthritis, grade 1 = doubtful joint space narrowing and possible osteophytic lipping, grade 2 = definite osteophytes and possible joint space narrowing).

Knee pain, functionality and force will be measured using validated measurement instruments. Pain and functionality will be our primary outcomes. Maximum, minimum and current pain intensity will be indicated on a 0-100 mm VAS line. Functionality will be measured using the Dutch version of the anterior knee pain scale (AKPS). The AKPS questionnaire consists of 13 items assessing subjective symptoms and functional limitations totalling a maximum score of 100. Our secondary outcome, maximum voluntary peak force (MVPF) of the quadriceps, will be measured using a Biodex system 3 isokinetic dynamometer (Biodex Medical Systems, Inc., Shirley, NY, USA). This system has shown sufficient reliability and validity for position, torque and velocity measurements in clinical and research settings. Patients will be assessed before intervention (=baseline), at 6 weeks (=immediately after the last intervention) and at 12 weeks (=6 weeks after the last intervention).

ELIGIBILITY:
Inclusion Criteria:

* self-reported unilateral or
* bilateral anterior knee pain provoked by at least two of the following activities: jumping, squatting, ascending/ descending stairs, kneeling, prolonged sitting and or a
* positive patellar compression test

Exclusion Criteria:

* experiencing pain for less than 3 months
* a history of knee surgery
* meniscal lesion
* patellar subluxation/dislocation
* evidence of tendinopathy or ligamentous pathologies
* dislocation or fracture in the pelvic region
* spinal surgery
* osteoporosis
* pregnancy
* neurologic disorders
* findings of chondromalacia > grade 2 on MRI, echography or X-ray.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2021-01-28 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | before the first intervention (at baseline)
  Maximum, minimum and current pain intensity was indicated on a 0-100 mm VAS line.
Visual analogue scale | 6 weeks after the first intervention (at 6 weeks)
  Maximum, minimum and current pain intensity was indicated on a 0-100 mm VAS line.
Visual analogue scale | 6 weeks after the last intervention (at 12 weeks)
  Maximum, minimum and current pain intensity was indicated on a 0-100 mm VAS line.
Functionality | before the first intervention (baseline)
  Functionality will be measured using the Dutch version of the anterior knee pain scale (AKPS). The AKPS questionnaire consists of 13 items assessing subjective symptoms and functional limitations totalling a maximum score of 100
Functionality | 6 weeks after the first intervention (at 6 weeks)
  Functionality will be measured using the Dutch version of the anterior knee pain scale (AKPS). The AKPS questionnaire consists of 13 items assessing subjective symptoms and functional limitations totalling a maximum score of 100
Functionality | 6 weeks after the last intervention (at 12 weeks)
  Functionality will be measured using the Dutch version of the anterior knee pain scale (AKPS). The AKPS questionnaire consists of 13 items assessing subjective symptoms and functional limitations totalling a maximum score of 100

SECONDARY OUTCOMES:
Knee extension strength | before the first intervention (baseline)
  Maximum voluntary peak force (MVPF) of the quadriceps, will be measured using a Biodex system 3 isokinetic dynamometer (Biodex Medical Systems, Inc., Shirley, NY, USA). This system has shown sufficient reliability and validity for position, torque and velocity measurements in clinical and research settings.
Knee extension strength | 6 weeks after the first intervention (at 6 weeks)
  Maximum voluntary peak force (MVPF) of the quadriceps, will be measured using a Biodex system 3 isokinetic dynamometer (Biodex Medical Systems, Inc., Shirley, NY, USA). This system has shown sufficient reliability and validity for position, torque and velocity measurements in clinical and research settings.
Knee extension strength | 6 weeks after the last intervention (at 12 weeks)
  Maximum voluntary peak force (MVPF) of the quadriceps, will be measured using a Biodex system 3 isokinetic dynamometer (Biodex Medical Systems, Inc., Shirley, NY, USA). This system has shown sufficient reliability and validity for position, torque and velocity measurements in clinical and research settings.

OTHER OUTCOMES:
Age | before intervention (at baseline)
  self-reported age (in years)
Weight | before intervention (at baseline)
  self-reported weight (in kg)
Height | before intervention (at baseline)
  self-reported height (in cm)
Duration of symptoms | before intervention (at baseline)
  self-reported duration of symptoms (in months)
Sport | before intervention (at baseline)
  self-reported weekly participation in sport (Yes/No)
Previous exercise therapy | before intervention (at baseline)
  self-reported previous exercise therapy treatment for the knee (Yes/No).
Chondral lesion | before intervention (at baseline)
  Grade of patellofemoral chondral lesion (Grade 0, Grade 1, Grade 2) using Kellgren and Lawrence system for classification of osteoarthritis (X-ray)

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Scafoglieri, Professor, Study Chair — Vrije Universiteit Brussel

IPD SHARING:
Plan to Share IPD: No
According to GDPR regulations upon reasonable request study results can be shared

REFERENCES:
- [Result] Fredericson M, Yoon K. Physical examination and patellofemoral pain syndrome. Am J Phys Med Rehabil. 2006 Mar;85(3):234-43. doi: 10.1097/01.phm.0000200390.67408.f0. PMID 16505640
- [Result] Suter E, McMorland G, Herzog W, Bray R. Decrease in quadriceps inhibition after sacroiliac joint manipulation in patients with anterior knee pain. J Manipulative Physiol Ther. 1999 Mar-Apr;22(3):149-53. doi: 10.1016/S0161-4754(99)70128-4. PMID 10220713
- [Result] Sueki DG, Cleland JA, Wainner RS. A regional interdependence model of musculoskeletal dysfunction: research, mechanisms, and clinical implications. J Man Manip Ther. 2013 May;21(2):90-102. doi: 10.1179/2042618612Y.0000000027. PMID 24421619
- [Result] Wainner RS, Whitman JM, Cleland JA, Flynn TW. Regional interdependence: a musculoskeletal examination model whose time has come. J Orthop Sports Phys Ther. 2007 Nov;37(11):658-60. doi: 10.2519/jospt.2007.0110. No abstract available. PMID 18057674
- [Result] Kooiker L, Van De Port IG, Weir A, Moen MH. Effects of physical therapist-guided quadriceps-strengthening exercises for the treatment of patellofemoral pain syndrome: a systematic review. J Orthop Sports Phys Ther. 2014 Jun;44(6):391-402, B1. doi: 10.2519/jospt.2014.4127. Epub 2014 Apr 25. PMID 24766358
- [Result] Hillermann B, Gomes AN, Korporaal C, Jackson D. A pilot study comparing the effects of spinal manipulative therapy with those of extra-spinal manipulative therapy on quadriceps muscle strength. J Manipulative Physiol Ther. 2006 Feb;29(2):145-9. doi: 10.1016/j.jmpt.2005.12.003. PMID 16461174
- [Result] Drouin JM, Valovich-mcLeod TC, Shultz SJ, Gansneder BM, Perrin DH. Reliability and validity of the Biodex system 3 pro isokinetic dynamometer velocity, torque and position measurements. Eur J Appl Physiol. 2004 Jan;91(1):22-9. doi: 10.1007/s00421-003-0933-0. Epub 2003 Sep 24. PMID 14508689
- [Result] Almosnino S, Stevenson JM, Bardana DD, Diaconescu ED, Dvir Z. Reproducibility of isokinetic knee eccentric and concentric strength indices in asymptomatic young adults. Phys Ther Sport. 2012 Aug;13(3):156-62. doi: 10.1016/j.ptsp.2011.09.002. Epub 2011 Oct 22. PMID 22814449
- [Derived] Scafoglieri A, Van den Broeck J, Willems S, Tamminga R, van der Hoeven H, Engelsma Y, Haverkamp S. Effectiveness of local exercise therapy versus spinal manual therapy in patients with patellofemoral pain syndrome: medium term follow-up results of a randomized controlled trial. BMC Musculoskelet Disord. 2021 May 15;22(1):446. doi: 10.1186/s12891-021-04310-9. PMID 33992100
- Available data/document: Individual Participant Data Set — https://vub-my.sharepoint.com/:f:/g/personal/aldo_scafoglieri_vub_be/EspOeK0bPk9JgvUpkobVcZEB-fPjar_48PO4_aIq-JhsIw?e=Wsu4DC — Access can be granted by the participant data set holder: Prof dr Aldo Scafoglieri